CLINICAL TRIAL: NCT04859894
Title: Lung Function, Heart Function and Aerobic Capacity in Patients Suffering From Long-term Symptoms Following SARS-CoV2-infection, and the Association With DNA Methylation
Brief Title: Physiological Studies in Post-COVID-19 Syndrome, and the Association With DNA Methylation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Kristofer Hedman, Associate Professor, Linkoeping University
Other Study IDs: 2021-01620
Record Dates: First submitted 2021-04-13; First posted 2021-04-26 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Cardiopulmonary Disease; Dyspnea; Lung Function Decreased; Epigenetic Disorder
Keywords: Cardiopulmonary Exercise Testing; Lung Function Testing; Echocardiography; DNA-methylation; Covid19
MeSH Terms: conditions — COVID-19; Pulmonary Heart Disease; Dyspnea; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum Venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid19: Patients aged >18 years with confirmed Covid19 disease with symptoms >12 weeks, not better explained by other disease
  Interventions: Diagnostic Test: Physiological testing

INTERVENTIONS:
Diagnostic Test: Physiological testing — Cardiopulmonary exercise testing, Lung Function Testing and in some cases echocardiography. 20 subjects will perform DNA-methylation testing.

SUMMARY:
The physiological derangements in subjects suffering from long-term symptoms following a Covid-19 infection (Post-COVID-19 Syndrome) are poorly understood and evaluated. This study will recruit subjects with a clinical diagnosis of Post-Covid-19-syndrome) who are scheduled for either of lung function testing, cardiopulmonary exercise testing or cardiac ultrasound. Patients' symptoms will be correlated to physiological measures and compared to predicted values. In addition, in 20 patients, symptoms and physiological measures will be correlated to epigenetical alterations, or DNA-methylation patterns. In addition, a subset of patients will be examined a year after the baseline testing in order to follow the progress of the disease.

DETAILED DESCRIPTION:
The physiological derangements in subjects suffering from long-term symptoms following a Covid-19 infection (Post-COVID-19 Syndrome) are poorly understood and evaluated. For example, the extent to which subjective symptoms correlate with physiological impairments are not known.

This study will recruit subjects with a clinical diagnosis of Post-Covid-19-syndrome) who are scheduled for either of lung function testing, cardiopulmonary exercise testing or cardiac ultrasound. Patients' symptoms will be correlated to physiological measures and compared to predicted values.

In addition, in 20 patients, symptoms and physiological measures will be correlated to epigenetical alterations, or DNA-methylation patterns. In addition, a subset of patients will be examined a year after the baseline testing in order to follow the progress of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or clinically highly suspected Covid19-infection
* Symptom duration at least 12 weeks following first occurence of symptoms
* No other disease that better could explain the symptoms than Covid19

Exclusion Criteria:

* Age <18 years
* Unability to perform a maximal exercise test
* Unability to understand written or spoken Swedish

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All subjects fulfilling inclusion criteria and no exclusion criterion referred for a clinical examination at the specified clinic will be informed about the study and inquired regarding participation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Peak Oxygen Consumption (VO2peak) | At baseline
  Cross-sectional evaluation of VO2peak and the association with symptoms

SECONDARY OUTCOMES:
Peak Oxygen Consumption (VO2peak) | In subset of subjects at 1 year
  Improvement in VO2peak over 1 year
VE/VCO2-slope | At baseline, in subset at 1 year
  Cross-sectional evaluation of VE/VCO2 and the association with symptoms
Diffusion Capacity (DLCOc) | At baseline, in subset at 1 year
  Cross-sectional evaluation of DLCOc and the association with symptoms
Forced Expiratory Volume in 1 second (FEV1) | At baseline, in subset at 1 year
  Cross-sectional evaluation of FEV1 and the association with symptoms
Forced Vital Capacity (FVC) | At baseline, in subset at 1 year
  Cross-sectional evaluation of FVC and the association with symptoms
Total Lung Capacity (TLC) | At baseline, in subset at 1 year
  Cross-sectional evaluation of TLC and the association with symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Dept Health, Medicine and Caring Sciences, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
As part of a national collaboration on Post Covid19, coded (deidentified) data may be shared with other selected researchers in accordance with the ethical permission obtained by the Ethical Review Board.